CLINICAL TRIAL: NCT02812641
Title: A Randomized Trial of Adding Bevacizumab to Neoadjuvant Platinum-Fluorouracil Concurrent Chemoradiation in Locally Advanced Esophageal Squamous Cell Carcinoma
Brief Title: Neoadjuvant CCRT With/Without Bevacizumab for Locally Advanced ESCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 201511008MINC
Record Dates: First submitted 2016-06-13; First posted 2016-06-24 (Estimated); Last update posted 2019-03-11 (Actual); Status verified 2019-03

CONDITIONS: Stage III Esophageal Squamous Cell Carcinoma
Keywords: Concurrent chemoradiation; Esophageal squamous cell carcinoma; Vascular endothelial growth factor
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Bevacizumab; Cisplatin; Fluorouracil; Radiation; Random Allocation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- BPF-CCRT (Run-in Phase) (Experimental): Neoadjuvant CCRT with Bevacizumab, Cisplatin and 5-fluorouracil
  Chemotherapy:
  Bevacizumab(B): 10 mg/kg on day 1
  Cisplatin(P): 75 mg/m2 on day 1
  5-fluorouracil(F): 24 hours continuous infusion of 1,000 mg/m2 on days 1-4
  Radiotherapy: 40 Gy/20 fractions: days 1-5, weeks 1-4
  Interventions: Drug: BPF-CCRT (run-in)
- BPF-CCRT (Randomized Phase) (Experimental): Neoadjuvant CCRT with Bevacizumab, Cisplatin and 5-fluorouracil
  Chemotherapy:
  Bevacizumab(B): 10 mg/kg on day 1
  Cisplatin(P): 75 mg/m2 on day 1
  5-fluorouracil(F): 24 hours continuous infusion of 1,000 mg/m2 on days 1-4
  Radiotherapy: 40 Gy/20 fractions: days 1-5, weeks 1-4
  Interventions: Drug: BPF-CCRT (randomized)
- PF-CCRT (Randomized Phase) (Active Comparator): Neoadjuvant CCRT with Cisplatin and 5-fluorouracil
  Chemotherapy:
  Cisplatin(P): 75 mg/m2 on day 1
  5-fluorouracil(F): 24 hours continuous infusion of 1,000 mg/m2 on days 1-4
  Radiotherapy: 40 Gy/20 fractions: days 1-5, weeks 1-4
  Interventions: Drug: PF-CCRT (randomized)

INTERVENTIONS:
Drug: BPF-CCRT (run-in) — Six patients will be enrolled in run-in phase. If <= 1 patient developed dose-limiting toxicity, the trial will be continued to randomized phase. If > 1 patients developed dose-limiting toxicities, the protocol will be discontinued.
  Other Names: Bevacizumab; Cisplatin; 5-Fluorouracil; Radiation
  Arms: BPF-CCRT (Run-in Phase)
Drug: BPF-CCRT (randomized) — Twenty-two patients will be planned to assign to the experimental arm
  Other Names: Bevacizumab; Cisplatin; 5-Fluorouracil; Radiation
  Arms: BPF-CCRT (Randomized Phase)
Drug: PF-CCRT (randomized) — Twenty-two patients will be planned to assign to the active control arm
  Other Names: Cisplatin; 5-Fluorouracil; Radiation
  Arms: PF-CCRT (Randomized Phase)

SUMMARY:
Esophageal squamous cell carcinoma (ESCC) is one of the ten leading cancers in Taiwanese male. The prognosis is poor with a five-year overall survival rate of 10 to 30 %. Randomized clinical trials have demonstrated that trimodality therapy (TMT), consisted of neoadjuvant concurrent chemoradiation (CCRT) and radical esophagectomy, improves the overall survival for patients with locally advanced disease. Despite of the advancement, the outcome remained unsatisfactory with the median progression-free survival around 20 to 25 months and median overall survival around 30 months. It is know that the most important prognostic factor is whether a pathological complete response can be achieved after neoadjuvant CCRT. However, the use of new generation chemotherapeutic agent taxanes and epidermal growth factor inhibitors (such as Cetuximab) failed to significantly improve prognosis comparing to the standard platinum-fluorouracil (PF) regimen. As a consequence, it is mandatory to develop new chemotherapeutic regimen for CCRT.

In previous prospective studies, investigators used proximal ligation assay technology to identify serum VEGF-A in correlation with the pathological response and prognosis for patients receiving neoadjuvant CCRT plus radical esophagectomy for locally advanced ESCC. Other investigators also showed high VEGF expression correlating to poor outcome. Therefore, investigators generate the hypothesis that adding vascular endothelial growth factor (VEGF) monoclonal antibody, Bevacizumab, to standard neoadjuvant CCRT may improve outcome for patients with ESCC. Meanwhile, several prospective clinical studies have shown the feasibility, safety, and activity of adding Bevacizumab to chemotherapy, CCRT, or combined modality therapy including surgery, either in head and neck cancer, esophageal cancer, or esophagogastric junction adenocarcinoma. However, its efficacy should be further investigated in larger prospective trials and little is known about the activity and toxicity of Bevacizumab in ESCC due to small number of reported cases. In the present clinical trial, investigators plan to investigate whether incorporation of Bevacizumab into standard neoadjuvant PF-CCRT will improve treatment response and increase pathological complete response rate. Investigators will also evaluate associated biomarkers in relation to prognosis. By the present research, investigators expect to develop a new TMT regimen for this poor prognostic disease.

DETAILED DESCRIPTION:
This study is a randomized trial to compare the outcomes between patients receiving neoadjuvant PF-CCRT plus Bevacizumab (BPF-CCRT) or PF-CCRT alone. Investigators design to enrol 6 patients in the run-in phase, and 44 patients in the randomized phase (22 patients in each group) to develop the preliminary evidence for using Bevacizumab in ESCC.

ELIGIBILITY:
Inclusion criteria

To be eligible for inclusion, patients must fulfill the following criteria:

1. Histologically proved squamous cell carcinoma of esophagus
2. Locoregional advanced stage III disease, which are defined by Tumor, Nodes, Metastases (TNM) system of American Joint Committee on Cancer (AJCC) Cancer Staging System (7th edition) in 2010, fulfilling one of the following criteria:

   1. T1-2 N2-3 M0
   2. T3 N1-3 M0
3. Medical fit for curative surgery
4. Age ≥ 20 years
5. Karnofsky Performance Status ≥ 60%
6. Adequate bone marrow reserves within 2 weeks prior to registration, defined as:

   1. white blood cells (WBC) ≥ 4,000/µl or neutrophil count (ANC) ≥ 2,000/µl
   2. platelets ≥ 100,000/µl
   3. hemoglobin ≥ 9.0 g/dl
7. Adequate liver function reserves within 2 weeks prior to registration, defined as:

   1. hepatic transaminases ≤ 2.5 x upper limit of normal (ULN)
   2. serum total bilirubin ≤ 1.5 x upper limit of normal (ULN)
8. Adequate renal function within 2 weeks prior to registration: Creatinine ≤1.5 mg/dL
9. International normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin time (aPTT) ≤ 1.5 X ULN within 2 weeks prior to registration
10. Women of childbearing potential and male participants must practice adequate contraception
11. Patients must be able to comply with the study protocol and follow-up schedules and provide study-specific informed consent

Exclusion criteria Patients fulfill any of the following criteria will be excluded from this trial

1. Prior radiotherapy to head and neck, chest, or abdomen
2. Tumor invasion to adjacent structures (T4 lesion)
3. Presence of distant metastasis
4. Adenocarcinoma of gastroesophageal junction.
5. Synchronously or metachronously diagnosed squamous cell carcinoma of aerodigestive way, other than oesophageal cancer
6. Prior invasive malignancy
7. Severe, active comorbidities which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and adverse events of the protocol, or limit compliance with study requirements, defined as follows:

   1. Uncontrolled active infection requiring intravenous antibiotics at the time of registration
   2. Transmural myocardial infarction ≤ 6 months prior to registration
   3. Unstable angina or congestive heart failure requiring hospitalization ≤ 6 months prior to registration
   4. Life-threatening uncontrolled clinically significant cardiac arrhythmias
   5. Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects
   6. Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of registration
   7. Uncontrolled psychiatric disorder
8. On full-dose anticoagulants (e.g., Warfarin or low molecular weight heparin) or medications known to inhibit platelet function (e.g. aspirin, dipyramidole, ticlopidine, clopidogrel, cilostazol, or NSAIDs)
9. Prior history of hypertensive crisis or blood pressure at baseline > 150/100 mmHg
10. Hepatic insufficiency resulting in coagulation defects
11. History of a non-healing wound, ulcer, or bone fracture within 90 days (3 months) prior to registration
12. Any hemorrhage/bleeding event CTCAE, ver. 4 grade 3 or greater within 30 days prior to registration
13. Gross hemoptysis or hematemesis (defined as bright red blood of 1 teaspoon or more or frank clots within minimal or no phlegm per coughing episode) within 4 weeks prior to registration; patients with incidental blood mixed with phlegm are not excluded.
14. Major surgical procedure or significant traumatic injury within 28 days prior to registration (with the exception of jejunostomy or port-A insertion)
15. Women of childbearing potential and male participants who are sexually active and not willing/able to use medically acceptable forms of contraception; this exclusion is necessary because the radiation treatment involved in this study may be significantly teratogenic

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2016-06; Primary Completion 2019-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting toxicity (run-in phase) | 30 days after radical esophagectomy
  Number of participant in the run-in phase with life-threatening adverse event or death, which is probable or definitely associated with bevacizumab
Pathological complete response rate (randomized phase) | 8 weeks
  Number of participant achieved pathological complete response, which is defined as complete surgical resection of all gross tumours without residual microscopic invasive carcinoma at primary tumor location and dissected lymph nodes.

SECONDARY OUTCOMES:
Acute toxicity | From date of CCRT until 90 days after CCRT starts
  Common Toxicity Criteria for Adverse Events version 4
Late toxicity | From 90 days after CCRT starts until the date of death from any cause, up to 60 months
  Common Toxicity Criteria for Adverse Events version 4
Patient reported outcome (Quality of Life questionnaire of cancer patients) | At baseline, 2, 4 weeks after CCRT, before surgery, 1 month after surgery, and every 3 month thereafter until unequivocal progression, hospice care, or death, assessed up to 24 months
  EORTC Quality of Life-Core 30 questionnaire module
Patient reported outcome (Quality of Life questionnaire of esophageal cancer patients) | At baseline, 2, 4 weeks after CCRT, before surgery, 1 month after surgery, and every 3 month thereafter until unequivocal progression, hospice care, or death, assessed up to 24 months
  EORTC Quality of Life-Oesophagus(OES) 18 questionnaire module
Image response | at baseline and before surgery (8 weeks)
  Response Evaluation Criteria In Solid Tumors version 1.1
Metabolic Image response | at baseline and before surgery (8 weeks)
  Positron Emission Tomography Response Criteria in Solid Tumors version 1.0
Progression-free survival | From date of enrolment until the date of first documented disease progression or date of death from any cause, whichever came first, assessed up to 60 months
  Number of participant with disease progression
Overall survival | From date of enrollment until the date of death from any cause, assessed up to 60 months
  Number of participant alive

OTHER OUTCOMES:
Serum biomarker (VEGF-A) | At baseline, after CCRT, before and after surgery, and documented disease progression, assessed up to 100 months
  Serum VEGF-A concentration measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Jason Chia-Hsien Cheng, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No